CLINICAL TRIAL: NCT00544583
Title: Continuous Versus Interrupted Abdominal Wall Closure After Emergency Midline Laparotomy: CONTINT - A Randomized Controlled Study
Brief Title: Continuous Versus Interrupted Abdominal Wall Closure After Emergency Midline Laparotomy
Acronym: CONTINT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: University of Heidelberg, Germany, Department of General, Visceral and Transplantation Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S206/2007
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Laparotomy; Hernia
Keywords: Abdominal wall
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Interrupted closure with Vicryl equivalent sutures (USP 2, 45 cm)
  Interventions: Procedure: Interrupted sutures
- B (Experimental): Continuous closure with PDS II equivalent sutures (USP 1, 150 cm loops)
  Interventions: Procedure: Continuous sutures

INTERVENTIONS:
Procedure: Interrupted sutures — Interrupted sutures for abdominal fascia closure with Vicryl equivalent sutures (USP 2, 45 cm)
  Arms: A
Procedure: Continuous sutures — Continuous sutures for abdominal fascia closure with PDS II equivalent USP 1, 150 cm loops
  Arms: B

SUMMARY:
Patients undergoing primary midline laparotomy for an emergency surgical intervention with a suspected septic focus in the abdominal cavity.

DETAILED DESCRIPTION:
More than 700.000 open abdominal surgeries (laparotomies) are performed each year in Germany (2). A major surgical complication after laparotomy is abdominal fascia dehiscence which might appear either as early (burst abdomen with evisceration) or as late complication (incisional hernia). These patients usually undergo surgery for secondary fascial closure associated with markedly increased morbidity (3) including high recurrence rates (up to 45%) (4). The applied surgical strategy of abdominal wall closure (i.e. the combination of suture technique and material) is of high relevance for prevention of fascia dehiscence and, moreover, constitutes the main factor directly controllable by the surgeon. While several randomized controlled trials (RCT) (3; 5-8) as well as meta-analyses (9-12) exist that address the issue of optimal fascia closure in elective laparotomies, there is no RCT dealing exclusively with the emergency setting. As a result abdominal fascia closure is performed according to the surgeon's individual preference rather than according to evidence-based data. Therefore, the present RCT is designed to compare the most established strategies (continuous slowly absorbable sutures and interrupted rapidly absorbable sutures) for abdominal wall closure in order to determine differences between both strategies after midline incisions.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative Inclusion criteria:

   * Age equal or greater than 18 years
   * Expected survival time more than 12 months
   * Patients undergoing primary and emergency midline laparotomy (patients with prior laparoscopy (not colon resections) or minor abdominal operation (e.g. appendectomy, cholecystectomy, hysterectomy, sectio) may be included into the trial)
   * Suspected septic abdominal focus (e.g. perforated stomach ulcer, perforated diverticulitis)
   * Informed consent
2. Intraoperative inclusion criteria before closure:

   * Successful source control
   * Abdominal lavage

Exclusion Criteria:

1. Preoperative exclusion criteria:

   * Participation in another intervention-trial with interference of intervention and outcome of this study
2. Intraoperative exclusion criteria before closure:

   * Planned re-laparotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-11; Primary Completion 2011-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia or burst abdomen within 12 months | 12 months

SECONDARY OUTCOMES:
Quality of Life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nuh N Rahbari, MD, Study Director — Department of Surgery, University of Heidelberg; Markus W Büchler, MD, Principal Investigator — Department of Surgery, University of Heidelberg
Locations (1):
- Department of Surgery, Heidelberg, Germany

REFERENCES:
- [Derived] Rahbari NN, Knebel P, Kieser M, Bruckner T, Bartsch DK, Friess H, Mihaljevic AL, Stern J, Diener MK, Voss S, Rossion I, Buchler MW, Seiler CM. Design and current status of CONTINT: continuous versus interrupted abdominal wall closure after emergency midline laparotomy - a randomized controlled multicenter trial [NCT00544583]. Trials. 2012 May 30;13:72. doi: 10.1186/1745-6215-13-72. PMID 22647387